CLINICAL TRIAL: NCT01449331
Title: Qualitative Outcomes After Palliative Noninvasive Mechanical Ventilation : OVNI Study
Brief Title: The Use of Palliative Non Invasive Ventilation in Acute Respiratory Failure. OVNI Study.
Acronym: OVNI
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM 09006
Record Dates: First submitted 2011-10-05; First posted 2011-10-10 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2012-11

CONDITIONS: Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is:

* to estimate the frequency of the use of non invasive ventilation
* to estimate the frequency of the use of palliative non invasive ventilation
* to evaluate the impact of non invasive ventilation
* to propose some recommendations

DETAILED DESCRIPTION:
The purpose of this study is:

* to estimate the frequency of the use of non invasive ventilation
* to estimate the frequency of the use of palliative non invasive ventilation
* to evaluate the impact
* to propose some recommendations

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure
* hospitalization in ICU
* age >= 18 years

Exclusion Criteria:

* Patients who have already participated to OVNI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non invasive ventilation in ICU
Sampling Method: Probability Sample
Enrollment: 1450 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Quality of life of patients receiving palliative noninvasive mechanical ventilation | day 90
  Quality of life, assessed by short-form (SF)-36 health survey at day 90 after ICU discharge (average expected duration=7 days)

SECONDARY OUTCOMES:
Anxiety and Depression (evaluated by HADS) | day 90
  Anxiety and depression at day 90 after ICU discharge (expected average duration=7 days), evaluated by Hospital Anxiety Depression Scale
Survival status | patients will be followed during an average time of 14 days (mean hospitalization time) and until day 90 after ICU discharge
  Survival status (0=alive, 1=deceased)at ICU discharge (average expected duration=7 days)and hospital discharge (average expected duration=14 days), day 90 after ICU discharge, day 180 after ICU discharge and 1 year after ICU discharge
Post traumatic stress disorder, evaluated by Impact of Event Scale(IES) questionnaire | day 90
  PTSD evaluated by the Impact of Event Scale at day 90 after ICU discharge (average expected duration=7 days)

CONTACTS AND LOCATIONS:
Overall Officials: Elie Azoulay, MD,PhD, Principal Investigator — Service de Réanimation Médicale, Hôpital Saint Louis, AP-HP, France
Locations (1):
- Hôpital Saint-Louis, AP-HP, Paris, France

REFERENCES:
- [Result] Demoule A, Chevret S, Carlucci A, Kouatchet A, Jaber S, Meziani F, Schmidt M, Schnell D, Clergue C, Aboab J, Rabbat A, Eon B, Guerin C, Georges H, Zuber B, Dellamonica J, Das V, Cousson J, Perez D, Brochard L, Azoulay E; oVNI Study Group; REVA Network (Research Network in Mechanical Ventilation). Changing use of noninvasive ventilation in critically ill patients: trends over 15 years in francophone countries. Intensive Care Med. 2016 Jan;42(1):82-92. doi: 10.1007/s00134-015-4087-4. Epub 2015 Oct 13. PMID 26464393
- [Result] Azoulay E, Kouatchet A, Jaber S, Lambert J, Meziani F, Schmidt M, Schnell D, Mortaza S, Conseil M, Tchenio X, Herbecq P, Andrivet P, Guerot E, Lafabrie A, Perbet S, Camous L, Janssen-Langenstein R, Collet F, Messika J, Legriel S, Fabre X, Guisset O, Touati S, Kilani S, Alves M, Mercat A, Similowski T, Papazian L, Meert AP, Chevret S, Schlemmer B, Brochard L, Demoule A. Noninvasive mechanical ventilation in patients having declined tracheal intubation. Intensive Care Med. 2013 Feb;39(2):292-301. doi: 10.1007/s00134-012-2746-2. Epub 2012 Nov 27. PMID 23184037
- [Derived] Dangers L, Montlahuc C, Kouatchet A, Jaber S, Meziani F, Perbet S, Similowski T, Resche-Rigon M, Azoulay E, Demoule A; REVA Network (Research Network in Mechanical Ventilation) and the Groupe de Recherche en Reanimation Respiratoire en Onco-Hematologie (GrrrOH); List of contributors who included study patients: Angers University Hospital, Angers, France:. Dyspnoea in patients receiving noninvasive ventilation for acute respiratory failure: prevalence, risk factors and prognostic impact: A prospective observational study. Eur Respir J. 2018 Aug 9;52(2):1702637. doi: 10.1183/13993003.02637-2017. Print 2018 Aug. PMID 29976650